CLINICAL TRIAL: NCT03128359
Title: A Pilot Study of Post-transplant High Dose Cyclophosphamide (PTCY) as Part of Graft-Versus-Host Disease (GVHD) Prophylaxis in T-Cell Replete HLA-Mismatched Unrelated Donor (MMUD) Ablative and Reduced Intensity Hematopoietic Cell Transplantation (HCT) for Hematological Malignancies
Brief Title: High Dose Cyclophosphamide, Tacrolimus, and Mycophenolate Mofetil in Preventing Graft Versus Host Disease in Patients With Hematological Malignancies Undergoing Myeloablative or Reduced Intensity Donor Stem Cell Transplant
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 16419; NCI-2017-00480 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 16419 (Other: City of Hope Medical Center)
Record Dates: First submitted 2017-03-24; First posted 2017-04-25 (Actual); Results first posted 2023-06-09 (Actual); Last update posted 2024-01-09 (Actual); Status verified 2024-01

CONDITIONS: Acute Leukemia; Chronic Lymphocytic Leukemia/Small Lymphocytic Lymphoma; Chronic Myelogenous Leukemia, BCR-ABL1 Positive; Diffuse Large B-Cell Lymphoma; Follicular Lymphoma; Graft Versus Host Disease; Hodgkin Lymphoma; Mantle Cell Lymphoma; Marginal Zone Lymphoma; Myelodysplastic Syndrome; Myeloproliferative Neoplasm; Recurrent Acute Myeloid Leukemia With Myelodysplasia-Related Changes; Recurrent Plasma Cell Myeloma; Refractory Plasma Cell Myeloma; Secondary Myelodysplastic Syndrome
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Follicular; Graft vs Host Disease; Hodgkin Disease; Lymphoma, Mantle-Cell; Lymphoma, B-Cell, Marginal Zone; Myelodysplastic Syndromes; Myeloproliferative Disorders; Multiple Myeloma | interventions — Busulfan; Cyclophosphamide; fludarabine phosphate; Stem Cell Transplantation; Hematopoietic Stem Cell Transplantation; Melphalan; Mycophenolic Acid; Peripheral Blood Stem Cell Transplantation; Tacrolimus; Whole-Body Irradiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Regimen A (fludarabine, melphalan, PBSC HCT, GVHD prophylaxis) (Experimental): Patients receive fludarabine phosphate IV over 60 minutes on days -7 to -3 and melphalan hydrochloride IV over 20 minutes on day -2.
  Patients undergo PBSC HCT on day 0.
  Patients receive cyclophosphamide IV over 1-2 hours on days 3-4, mycophenolate mofetil IV or PO TID beginning on days 5 and stopping on day 35 if no severe GVHD is present-35, and tacrolimus IV continuously on days 5-180 with a taper beginning on day 90 in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Cyclophosphamide; Drug: Fludarabine Phosphate; Procedure: Hematopoietic Cell Transplantation; Other: Laboratory Biomarker Analysis; Drug: Melphalan Hydrochloride; Drug: Mycophenolate Mofetil; Procedure: Peripheral Blood Stem Cell Transplantation; Other: Quality-of-Life Assessment; Drug: Tacrolimus
- Regimen B (fludarabine, busulfan, PBSC HCT, GVHD prophylaxis) (Experimental): Patients receive fludarabine phosphate IV over 1-3 hours and busulfan IV over 3 hour on days -5 to -2.
  Patients undergo PBSC HCT on day 0.
  Patients receive cyclophosphamide IV over 1-2 hours on days 3-4, mycophenolate mofetil IV or PO TID beginning on days 5 and stopping on day 35 if no severe GVHD is present-35, and tacrolimus IV continuously on days 5-180 with a taper beginning on day 90 in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Busulfan; Drug: Cyclophosphamide; Drug: Fludarabine Phosphate; Procedure: Hematopoietic Cell Transplantation; Other: Laboratory Biomarker Analysis; Drug: Mycophenolate Mofetil; Procedure: Peripheral Blood Stem Cell Transplantation; Other: Quality-of-Life Assessment; Drug: Tacrolimus
- Regimen C (fludarabine, TBI, PBSC HCT, GVHD prophylaxis) (Experimental): Patients receive fludarabine phosphate IV over 60 minutes on days -7 to -5 and TBI BID on days -4 to -1.
  Patients undergo PBSC HCT on day 0.
  Patients receive cyclophosphamide IV over 1-2 hours on days 3-4, mycophenolate mofetil IV or PO TID beginning on days 5 and stopping on day 35 if no severe GVHD is present-35, and tacrolimus IV continuously on days 5-180 with a taper beginning on day 90 in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Cyclophosphamide; Drug: Fludarabine Phosphate; Procedure: Hematopoietic Cell Transplantation; Other: Laboratory Biomarker Analysis; Drug: Mycophenolate Mofetil; Procedure: Peripheral Blood Stem Cell Transplantation; Other: Quality-of-Life Assessment; Drug: Tacrolimus; Radiation: Total-Body Irradiation

INTERVENTIONS:
Drug: Busulfan — Given IV
  Other Names: 1, 4-Bis[methanesulfonoxy]butane; BUS; Bussulfam; Busulfanum; Busulfex; Busulphan; CB 2041; CB-2041; Glyzophrol; GT 41; GT-41; Joacamine; Methanesulfonic Acid Tetramethylene Ester; Methanesulfonic acid, tetramethylene ester; Mielucin; Misulban; Misulfan; Mitosan; Myeleukon; Myeloleukon; Myelosan; Mylecytan; Myleran; Sulfabutin; Tetramethylene Bis(methanesulfonate); Tetramethylene bis[methanesulfonate]; WR-19508
  Arms: Regimen B (fludarabine, busulfan, PBSC HCT, GVHD prophylaxis)
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR- 138719
Drug: Fludarabine Phosphate — Given IV
  Other Names: 2-F-ara-AMP; 9H-Purin-6-amine, 2-fluoro-9-(5-O-phosphono-.beta.-D-arabinofuranosyl)-; Beneflur; Fludara; SH T 586
Procedure: Hematopoietic Cell Transplantation — Undergo PBSC HCT
  Other Names: HCT; Hematopoietic Stem Cell Transplantation; HSCT; stem cell transplantation
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Melphalan Hydrochloride — Given IV
  Other Names: Alkeran; Alkerana; Evomela
  Arms: Regimen A (fludarabine, melphalan, PBSC HCT, GVHD prophylaxis)
Drug: Mycophenolate Mofetil — Given IV or PO
  Other Names: Cellcept; MMF
Procedure: Peripheral Blood Stem Cell Transplantation — Undergo PBSC HCT
  Other Names: PBPC transplantation; Peripheral Blood Progenitor Cell Transplantation; Peripheral Stem Cell Support; Peripheral Stem Cell Transplant; Peripheral Stem Cell Transplantation
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Drug: Tacrolimus — Given IV
  Other Names: FK 506; Fujimycin; Hecoria; Prograf; Protopic
Radiation: Total-Body Irradiation — Undergo TBI
  Other Names: TOTAL BODY IRRADIATION; Whole-Body Irradiation
  Arms: Regimen C (fludarabine, TBI, PBSC HCT, GVHD prophylaxis)

SUMMARY:
This pilot phase II trial studies how well high dose cyclophosphamide, tacrolimus, and mycophenolate mofetil work in preventing graft versus host disease in patients with hematological malignancies undergoing myeloablative or reduced intensity donor stem cell transplant. Sometimes the transplanted cells from a donor can make an immune response against the body's normal cells (called graft versus host disease). Giving high dose cyclophosphamide, tacrolimus, and mycophenolate mofetil after the transplant may stop this from happening.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To estimate the graft versus host disease (GVHD)-free relapse/progression-free survival (GRFS) at one-year post hematopoietic cell transplantation (HCT) and to evaluate the clinical activity of post-transplant high dose cyclophosphamide (PTCy).

SECONDARY OBJECTIVES:

I. To summarize toxicities/complications/infections including type, frequency, severity, attribution, time course and duration through 100 days post-transplant.

II. To estimate the cumulative incidence (CI) of acute and chronic GVHD. III. To characterize the time course of neutrophil and platelet recovery/engraftment.

IV. To estimate overall survival (OS), progression-free survival (PFS), CI of relapse/progression and non-relapse mortality (NRM) at 100 days, 1 year and 2 years.

V. To describe quality of life at 100 days, 6 months, 1 and 2 years. VI. To characterize immune cell reconstitution and T cell repertoire post high dose cyclophosphamide in mismatched donor HCT.

VII. To characterize quality of life.

OUTLINE:

CONDITIONING REGIMEN: Patients are assigned to 1 of 3 conditioning regimens at the discretion of the attending physician and principal investigator.

REGIMEN A (REDUCED INTENSITY CONDITIONING): Patients receive fludarabine phosphate intravenously (IV) over 60 minutes on days -7 to -3 and melphalan hydrochloride IV over 20 minutes on day -2.

REGIMEN B (MYELOABLATIVE CONDITIONING [MAC]): Patients receive fludarabine phosphate IV over 1-3 hours and busulfan IV over 3 hour on days -5 to -2.

REGIMEN C (MAC): Patients receive fludarabine phosphate IV over 60 minutes on days -7 to -5 and total body irradiation (TBI) twice daily (BID) on days -4 to -1.

TRANSPLANT: Patients undergo peripheral blood stem cell (PBSC) hematopoietic cell transplantation (HCT) on day 0.

GVHD PROPHYLAXIS: Patients receive cyclophosphamide IV over 1-2 hours on days 3-4, mycophenolate mofetil IV or orally (PO) thrice daily (TID) beginning on day 5 and stopping on day 35 if no severe GVHD is present, and tacrolimus IV continuously on days 5-180 with a taper beginning on day 90 in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up twice weekly for 100 days, twice monthly for 6 months, monthly until no evidence of GVHD, and then yearly for up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients with acute leukemia or chronic myelogenous leukemia with no circulating blasts and with less than 10% blasts in the bone marrow
* Patients with myelodysplastic syndrome (MDS) with intermediate-2 or high risk per International Prognostic Scoring System (IPSS) (or intermediate, high, very high risk by Revised International Prognostic Scoring System [IPSS-R]) or myeloproliferative neoplasm; primary or secondary if high-risk features or refractory disease
* Patients with chronic lymphocytic leukemia/small lymphocytic lymphoma, follicular, marginal zone, diffuse large B-cell, Hodgkin lymphoma, or mantle cell lymphoma with chemosensitive disease at time of transplantation; all types of lymphoma are eligible
* High risk, or refractory and relapsed multiple myeloma
* No available human leukocyte antigen (HLA)-matched related donor
* Available matched unrelated donor
* Ejection fraction at rest >= 50%
* Karnofsky performance status (KPS) >= 70
* Measured creatinine clearance more than 60 mL/min. The updated Schwartz formula should be used for pediatric patients (>=5 to 12 years old)
* Carbon monoxide diffusing capability test (DLCO) >= 50% (adjusted for hemoglobin) and forced expiratory volume in 1 second (FEV1) >= 50%
* Total bilirubin < 1.5 x the upper limit of normal; patients who have been diagnosed with Gilbert's disease are allowed to exceed the defined bilirubin value of 1.5 x the upper limit of normal
* Alanine aminotransferase (ALT)/aspartate aminotransferase (AST) < 2.5 x the upper limit of normal
* Alkaline phosphatase < 2.5 x the upper limit of normal
* Female subjects (unless postmenopausal for at least 1 year before the screening visit, or surgically sterilized), agree to practice two (2) effective methods of contraception at the same time, or agree to completely abstain from heterosexual intercourse, from the time of signing of the informed consent through 12 months post-transplant
* Male subjects (even if surgically sterilized), of partners of women of childbearing potential must agree to one of the following: practice effective barrier contraception, or abstain from heterosexual intercourse from the time of signing the informed consent through 12 months post-transplant
* All subjects must have the ability to understand and the willingness to sign a written informed consent document

DONOR INCLUSION CRITERIA

* 7 out of 8 at high resolution using deoxyribonucleic acid (DNA)-based typing with either antigen or allele mismatched HLA (-A, -B, -C, and -DR) or 8/8 HLA-mismatched with either double DQ mismatch (10/12) or combined DQ and DP mismatch
* Donor must be willing to donate peripheral blood stem cells
* Suitable donor
* Medically cleared to donate per National Marrow Donor Program (NMDP)
* Absence of donor-specific antibodies (DSA) to the mismatched HLA-locus
* Donor choices per matched unrelated donor (MUD) committee according to center standard operating procedure (SOP)

Exclusion Criteria:

* Prior allogeneic transplant
* Active central nervous system (CNS) involvement by malignant cells
* Patients with uncontrolled bacterial, viral or fungal infections (currently taking medication and with progression or no clinical improvement) at time of enrollment
* Patients with transformed lymphoma (e.g., Richter's transformation arising in follicular lymphoma or chronic lymphocytic leukemia)
* Patients seropositive for the human immunodeficiency virus (HIV)
* Patients with active hepatitis B or C determined by polymerase chain reaction (PCR)
* Myocardial infarction within 6 months prior to enrollment or New York Heart Association (NYHA) class III or IV heart failure, uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities; prior to study entry, any electrocardiography (ECG) abnormality at screening must be documented by the investigator as not medically relevant
* Female patients who are lactating or pregnant
* Patients with a serious medical or psychiatric illness likely to interfere with participation in this clinical study
* History of another primary malignancy that has not been in remission for at least 3 years (the following are exempt from the 3-year limit: non-melanoma skin cancer, fully excised melanoma in situ [Stage 0], curatively treated localized prostate cancer, and cervical or breast carcinoma in situ on biopsy or a squamous intraepithelial lesion on PAP smear)
* Psychosocial issues: no appropriate caregivers identified, or non-compliant to medications
* Subjects, who in the opinion of the investigator, may not be able to comply with the safety monitoring requirements of the study

Ages: 5 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2017-05-30 (Actual); Primary Completion 2020-08-01 (Actual); Study Completion 2021-09-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Monzr Al Malki, MD, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States

REFERENCES:
- [Derived] Al Malki MM, Tsai NC, Palmer J, Mokhtari S, Tsai W, Cao T, Ali H, Salhotra A, Arslan S, Aldoss I, Karras N, Karanes C, Zain J, Khaled S, Stein A, Snyder D, Marcucci G, Forman SJ, Nakamura R. Posttransplant cyclophosphamide as GVHD prophylaxis for peripheral blood stem cell HLA-mismatched unrelated donor transplant. Blood Adv. 2021 Jun 22;5(12):2650-2659. doi: 10.1182/bloodadvances.2021004192. PMID 34156440

RESULTS

PARTICIPANT FLOW:
Groups:
- Regimen A (Fludarabine, Melphalan, PBSC HCT, GVHD Prophylaxis): Patients receive fludarabine phosphate IV over 60 minutes on days -7 to -3 and melphalan hydrochloride IV over 20 minutes on day -2.
  Patients undergo PBSC HCT on day 0.
  Patients receive cyclophosphamide IV over 1-2 hours on days 3-4, mycophenolate mofetil IV or PO TID beginning on days 5 and stopping on day 35 if no severe GVHD is present-35, and tacrolimus IV continuously on days 5-180 with a taper beginning on day 90 in the absence of disease progression or unacceptable toxicity.
  Cyclophosphamide: Given IV
  Fludarabine Phosphate: Given IV
  Hematopoietic Cell Transplantation: Undergo PBSC HCT
  Laboratory Biomarker Analysis: Correlative studies
  Melphalan Hydrochloride: Given IV
  Mycophenolate Mofetil: Given IV or PO
  Peripheral Blood Stem Cell Transplantation: Undergo PBSC HCT
  Quality-of-Life Assessment: Ancillary studies
  Tacrolimus: Given IV
- Regimen B (Fludarabine, Busulfan, PBSC HCT, GVHD Prophylaxis): Patients receive fludarabine phosphate IV over 1-3 hours and busulfan IV over 3 hour on days -5 to -2.
  Patients undergo PBSC HCT on day 0.
  Patients receive cyclophosphamide IV over 1-2 hours on days 3-4, mycophenolate mofetil IV or PO TID beginning on days 5 and stopping on day 35 if no severe GVHD is present-35, and tacrolimus IV continuously on days 5-180 with a taper beginning on day 90 in the absence of disease progression or unacceptable toxicity.
  Busulfan: Given IV
  Cyclophosphamide: Given IV
  Fludarabine Phosphate: Given IV
  Hematopoietic Cell Transplantation: Undergo PBSC HCT
  Laboratory Biomarker Analysis: Correlative studies
  Mycophenolate Mofetil: Given IV or PO
  Peripheral Blood Stem Cell Transplantation: Undergo PBSC HCT
  Quality-of-Life Assessment: Ancillary studies
  Tacrolimus: Given IV
- Regimen C (Fludarabine, TBI, PBSC HCT, GVHD Prophylaxis): Patients receive fludarabine phosphate IV over 60 minutes on days -7 to -5 and TBI BID on days -4 to -1.
  Patients undergo PBSC HCT on day 0.
  Patients receive cyclophosphamide IV over 1-2 hours on days 3-4, mycophenolate mofetil IV or PO TID beginning on days 5 and stopping on day 35 if no severe GVHD is present-35, and tacrolimus IV continuously on days 5-180 with a taper beginning on day 90 in the absence of disease progression or unacceptable toxicity.
  Cyclophosphamide: Given IV
  Fludarabine Phosphate: Given IV
  Hematopoietic Cell Transplantation: Undergo PBSC HCT
  Laboratory Biomarker Analysis: Correlative studies
  Mycophenolate Mofetil: Given IV or PO
  Peripheral Blood Stem Cell Transplantation: Undergo PBSC HCT
  Quality-of-Life Assessment: Ancillary studies
  Tacrolimus: Given IV
  Total-Body Irradiation: Undergo TBI
Period: Overall Study
Arm/Group | Regimen A (Fludarabine, Melphalan, PBSC HCT, GVHD Prophylaxis) | Regimen B (Fludarabine, Busulfan, PBSC HCT, GVHD Prophylaxis) | Regimen C (Fludarabine, TBI, PBSC HCT, GVHD Prophylaxis)
Started | 19 | 0 | 19
Completed | 19 | 0 | 19
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: No subject enrolled onto Regimen B.
Groups:
- Total: Total of all reporting groups
Arm/Group | Regimen A (Fludarabine, Melphalan, PBSC HCT, GVHD Prophylaxis) | Regimen B (Fludarabine, Busulfan, PBSC HCT, GVHD Prophylaxis) | Regimen C (Fludarabine, TBI, PBSC HCT, GVHD Prophylaxis) | Total
Number analyzed (Participants) | 19 | 0 | 19 | 38
Age, Continuous [Median (Full Range); unit: years] | 63 [33 to 72] |  | 44 [21 to 57] | 53 [21 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 |  | 11 | 19
  Male | 11 |  | 8 | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 |  | 8 | 11
  Not Hispanic or Latino | 15 |  | 11 | 26
  Unknown or Not Reported | 1 |  | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 |  | 0 | 0
  Asian | 4 |  | 4 | 8
  Native Hawaiian or Other Pacific Islander | 0 |  | 0 | 0
  Black or African American | 2 |  | 2 | 4
  White | 12 |  | 12 | 24
  More than one race | 0 |  | 0 | 0
  Unknown or Not Reported | 1 |  | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 19 |  | 19 | 38

OUTCOME MEASURES:

1. Primary Outcome: Graft-Versus-Host Disease-Free, Relapse-Free Survival (GRFS) at 1 Year
Description: Estimates will be calculated using the Kaplan-Meier method, Greenwood formula will be used to calculate standard error (SE), and log-log transformation method will be used to construct 95% confidence intervals. Graft versus host disease (GVHD, acute and chronic), disease status and vital status will be monitored per clinical standard operating procedure. For this endpoint failure is defined as the first occurrence of grade 3 or 4 acute GVHD, or moderate/severe chronic GVHD, or disease relapse (for patients in complete remission at the start of conditioning) or disease progression (for patients with active disease at the start of conditioning) or death (from any cause). Patients not experiencing any of these will be censored at his/her date of last contact.
Time Frame: From stem cell infusion to grade 3-4 acute graft versus host disease (GVHD), moderate-severe chronic GVHD, relapse, progression or death (from any cause), whichever occurs first, assessed for up to 1 year.
Measure: Number (95% Confidence Interval); unit: percentage of survival probability
Arm/Group | Regimen A (Fludarabine, Melphalan, PBSC HCT, GVHD Prophylaxis) | Regimen C (Fludarabine, TBI, PBSC HCT, GVHD Prophylaxis)
Number analyzed (Participants) | 19 | 19
percentage of survival probability | 53 [29 to 72] | 84 [59 to 95]

2. Secondary Outcome: Acute Graft Versus Host Disease (aGVHD) of Grades 2-4 According to the Consensus Grading
Description: Acute graft versus host disease is graded according to the 1994 Keystone Consensus Grading. aGVHD grade was evaluated from day 0 through 100 days post-transplant. The first day of acute GVHD onset at grades 2-4 was used to calculate the cumulative incidence. Relapse/death prior to onset was considered competing events.
Time Frame: Up to 100 days post-stem cell infusion
Measure: Number (95% Confidence Interval); unit: percentage of probability
Arm/Group | Regimen A (Fludarabine, Melphalan, PBSC HCT, GVHD Prophylaxis) | Regimen C (Fludarabine, TBI, PBSC HCT, GVHD Prophylaxis)
Number analyzed (Participants) | 19 | 19
percentage of probability | 47 [29 to 76] | 53 [34 to 81]

3. Secondary Outcome: Overall Survival (OS) at 1 Year
Description: Estimates was calculated using the Kaplan-Meier method, Greenwood formula was used to calculate SE, and log-log transformation method was used to construct 95% confidence intervals. Each patient's vital status was monitored per clinical standard operating procedure. For this endpoint failure is defined as death (from any cause). Patients not experiencing a death event was censored at his/her date of last contact.
Time Frame: From start of transplant to death, or last follow up, whichever occurs first, assessed for up to 1 year.
Measure: Number (95% Confidence Interval); unit: percentage of probability
Arm/Group | Regimen A (Fludarabine, Melphalan, PBSC HCT, GVHD Prophylaxis) | Regimen C (Fludarabine, TBI, PBSC HCT, GVHD Prophylaxis)
Number analyzed (Participants) | 19 | 19
percentage of probability | 68 [42 to 84] | 100 [NA to NA] — The 95% confidence intervals were not calculable because no participant reached the event at the final time point for assessment.

ADVERSE EVENTS:
Time Frame: Up to 2 years post-transplant.
Arm/Group | Regimen A (Fludarabine, Melphalan, PBSC HCT, GVHD Prophylaxis) | Regimen C (Fludarabine, TBI, PBSC HCT, GVHD Prophylaxis)
All-Cause Mortality (participants affected / at risk) | 9/19 | 0/19
Serious Adverse Events (participants affected / at risk) | 12/19 | 6/19
Other Adverse Events (participants affected / at risk) | 19/19 | 19/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Regimen A (Fludarabine, Melphalan, PBSC HCT, GVHD Prophylaxis) (N=19) | Regimen C (Fludarabine, TBI, PBSC HCT, GVHD Prophylaxis) (N=19)
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
HEMOLYSIS (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
ABDOMINAL PAIN (Gastrointestinal disorders) | 1 (1) | 0 (0)
DIARRHEA (Gastrointestinal disorders) | 1 (1) | 0 (0)
NAUSEA (Gastrointestinal disorders) | 0 (0) | 1 (1)
PANCREATITIS (Gastrointestinal disorders) | 0 (0) | 1 (1)
VOMITING (Gastrointestinal disorders) | 0 (0) | 2 (2)
CHILLS (General disorders) | 1 (1) | 1 (1)
FEVER (General disorders) | 0 (0) | 2 (2)
CMV VIREMIA (Infections and infestations) | 2 (2) | 0 (0)
ENTEROBACTER BACTEREMIA (Infections and infestations) | 1 (1) | 0 (0)
NOCARDIA INFECTION (Infections and infestations) | 1 (1) | 0 (0)
PNEUMONIA (Infections and infestations) | 1 (1) | 0 (0)
SEPSIS (Infections and infestations) | 3 (4) | 1 (1)
URINARY TRACT INFECTION (Infections and infestations) | 1 (1) | 0 (0)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 1 (1) | 0 (0)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 1 (1) | 0 (0)
CREATININE INCREASED (Investigations) | 1 (1) | 0 (0)
DISEASE RELAPSE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
RELAPSED DISEASE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
ADULT RESPIRATORY DISTRESS SYNDROME (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
DYSPNEA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Regimen A (Fludarabine, Melphalan, PBSC HCT, GVHD Prophylaxis) (N=19) | Regimen C (Fludarabine, TBI, PBSC HCT, GVHD Prophylaxis) (N=19)
ANEMIA (Blood and lymphatic system disorders) | 19 (43) | 19 (38)
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 17 (20) | 9 (9)
HEMOLYSIS (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
HEMOLYTIC UREMIC SYNDROME (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
LEFT NECK NODULE (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
LEUKOCYTOSIS (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
LYMPH NODE PAIN (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
ATRIAL FIBRILLATION (Cardiac disorders) | 1 (1) | 0 (0)
ATRIAL FLUTTER (Cardiac disorders) | 1 (1) | 0 (0)
ATRIOVENTRICULAR BLOCK FIRST DEGREE (Cardiac disorders) | 1 (1) | 0 (0)
CARDIOMEGALY (Cardiac disorders) | 1 (1) | 0 (0)
CHEST PAIN CARDIAC (Cardiac disorders) | 1 (1) | 0 (0)
GR DIASTOLIC DYSFUNCTION (Cardiac disorders) | 1 (1) | 0 (0)
HEART FAILURE (Cardiac disorders) | 1 (1) | 0 (0)
MYOCARDIAL INFARCTION (Cardiac disorders) | 1 (1) | 0 (0)
PALPITATIONS (Cardiac disorders) | 0 (0) | 1 (1)
PAROXYSMAL ATRIAL TACHYCARDIA (Cardiac disorders) | 1 (1) | 0 (0)
PERICARDIAL EFFUSION (Cardiac disorders) | 3 (3) | 0 (0)
RIGHT VENTRICULAR DYSFUNCTION (Cardiac disorders) | 1 (1) | 0 (0)
SINUS BRADYCARDIA (Cardiac disorders) | 2 (2) | 7 (9)
SINUS TACHYCARDIA (Cardiac disorders) | 17 (20) | 16 (21)
SR WITH PVCS (Cardiac disorders) | 1 (1) | 0 (0)
SUPRAVENTRICULAR TACHYCARDIA (Cardiac disorders) | 1 (1) | 0 (0)
EAR PAIN (Ear and labyrinth disorders) | 1 (1) | 1 (1)
TINNITUS (Ear and labyrinth disorders) | 1 (2) | 0 (0)
ADRENAL HYPERPLASIA (Endocrine disorders) | 1 (1) | 0 (0)
BLURRED VISION (Eye disorders) | 2 (3) | 2 (3)
CONJUNCTIVAL HEMORRHAGE (Eye disorders) | 1 (1) | 0 (0)
DRY EYE (Eye disorders) | 2 (2) | 2 (2)
FLASHING LIGHTS (Eye disorders) | 1 (1) | 0 (0)
FLOATERS (Eye disorders) | 0 (0) | 1 (2)
RT EYE IRRITATION (Eye disorders) | 1 (1) | 0 (0)
SUBCONJUNCTIVAL HEMORRHAGE (Eye disorders) | 1 (1) | 0 (0)
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 6 (6) | 0 (0)
ABDOMINAL PAIN (Gastrointestinal disorders) | 16 (19) | 13 (18)
ANAL HEMORRHAGE (Gastrointestinal disorders) | 1 (1) | 0 (0)
ANAL PAIN (Gastrointestinal disorders) | 0 (0) | 1 (1)
ASCITES (Gastrointestinal disorders) | 1 (1) | 0 (0)
BLOATING (Gastrointestinal disorders) | 1 (1) | 0 (0)
CHEILITIS (Gastrointestinal disorders) | 0 (0) | 1 (1)
COLITIS (Gastrointestinal disorders) | 2 (3) | 1 (1)
CONSTIPATION (Gastrointestinal disorders) | 6 (7) | 6 (10)
DENTAL CARIES (Gastrointestinal disorders) | 1 (1) | 1 (1)
DIARRHEA (Gastrointestinal disorders) | 19 (22) | 19 (20)
DRY MOUTH (Gastrointestinal disorders) | 13 (14) | 9 (11)
DUODENAL HEMORRHAGE (Gastrointestinal disorders) | 1 (1) | 0 (0)
DYSPEPSIA (Gastrointestinal disorders) | 5 (5) | 4 (4)
DYSPHAGIA (Gastrointestinal disorders) | 2 (3) | 6 (6)
FECAL INCONTINENCE (Gastrointestinal disorders) | 6 (6) | 1 (1)
FLATULENCE (Gastrointestinal disorders) | 2 (2) | 1 (1)
GASTRITIS (Gastrointestinal disorders) | 1 (1) | 0 (0)
GASTROESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 2 (2) | 4 (4)
GASTROPARESIS (Gastrointestinal disorders) | 1 (1) | 0 (0)
GINGIVAL PAIN (Gastrointestinal disorders) | 0 (0) | 1 (1)
HEMORRHOIDAL HEMORRHAGE (Gastrointestinal disorders) | 1 (1) | 0 (0)
HEMORRHOIDS (Gastrointestinal disorders) | 8 (8) | 5 (5)
ILEUS (Gastrointestinal disorders) | 1 (2) | 0 (0)
LOWER GASTROINTESTINAL HEMORRHAGE (Gastrointestinal disorders) | 1 (1) | 0 (0)
MUCOSITIS ORAL (Gastrointestinal disorders) | 13 (15) | 17 (18)
NAUSEA (Gastrointestinal disorders) | 19 (33) | 19 (30)
ORAL PAIN (Gastrointestinal disorders) | 3 (3) | 3 (3)
PERIANAL PAIN (Gastrointestinal disorders) | 0 (0) | 1 (1)
RECTAL HEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 1 (1)
RECTAL PAIN (Gastrointestinal disorders) | 6 (6) | 4 (4)
SALIVARY DUCT INFLAMMATION (Gastrointestinal disorders) | 0 (0) | 1 (1)
SMALL INTESTINAL MUCOSITIS (Gastrointestinal disorders) | 1 (1) | 0 (0)
VOMITING (Gastrointestinal disorders) | 18 (22) | 17 (25)
CHILLS (General disorders) | 11 (12) | 5 (5)
EDEMA FACE (General disorders) | 5 (5) | 1 (1)
EDEMA LIMBS (General disorders) | 15 (17) | 11 (13)
FATIGUE (General disorders) | 18 (21) | 18 (23)
FEVER (General disorders) | 16 (19) | 14 (14)
GAIT DISTURBANCE (General disorders) | 1 (2) | 0 (0)
HYPOTHERMIA (General disorders) | 1 (1) | 0 (0)
INFUSION RELATED REACTION (General disorders) | 4 (4) | 0 (0)
INJECTION SITE REACTION (General disorders) | 0 (0) | 2 (2)
IRRITABILITY (General disorders) | 0 (0) | 1 (1)
LOCALIZED EDEMA (General disorders) | 4 (4) | 1 (1)
MALAISE (General disorders) | 0 (0) | 1 (1)
NONCARDIAC CHEST PAIN (General disorders) | 5 (5) | 5 (5)
PAIN (General disorders) | 11 (18) | 6 (8)
CHOLELITHIASIS (Hepatobiliary disorders) | 1 (1) | 0 (0)
HEPATOMEGALY (Hepatobiliary disorders) | 1 (1) | 0 (0)
ALLERGIC REACTION (Immune system disorders) | 2 (2) | 0 (0)
CYTOKINE RELEASE SYNDROME (Immune system disorders) | 2 (2) | 1 (1)
ADENOVIRUS VIREMA (Infections and infestations) | 0 (0) | 1 (1)
BLADDER INFECTION (Infections and infestations) | 0 (0) | 1 (1)
CATHETER RELATED INFECTION (Infections and infestations) | 2 (2) | 2 (2)
CITROBACTER FREUNDII BACTEREMIA (Infections and infestations) | 0 (0) | 1 (1)
CMV (Infections and infestations) | 0 (0) | 1 (1)
CMV REACTIVATION (Infections and infestations) | 0 (0) | 1 (1)
CMV VIREMIA (Infections and infestations) | 0 (0) | 2 (2)
CORONAVIRUS (Infections and infestations) | 0 (0) | 1 (1)
E COLI BACTEREMIA (Infections and infestations) | 1 (1) | 1 (1)
ENTEROCOCCUS FAECALIS INFECTION (Infections and infestations) | 0 (0) | 1 (1)
ENTEROCOLITIS INFECTIOUS (Infections and infestations) | 1 (1) | 0 (0)
HERPES SIMPLEX (Infections and infestations) | 1 (1) | 0 (0)
HERPES VIRUS (Infections and infestations) | 1 (1) | 1 (1)
KLEBSIELLA PNEUMONIAIE (Infections and infestations) | 1 (1) | 0 (0)
LUNG INFECTION (Infections and infestations) | 2 (2) | 1 (1)
NAIL INFECTION (Infections and infestations) | 1 (1) | 0 (0)
POSITIVE CMV PCR (Infections and infestations) | 1 (1) | 0 (0)
S. VIRIDANS BACTEREMIA (Infections and infestations) | 0 (0) | 1 (1)
SEPSIS (Infections and infestations) | 1 (1) | 0 (0)
SINUSITIS (Infections and infestations) | 0 (0) | 1 (1)
SKIN INFECTION (Infections and infestations) | 2 (2) | 1 (1)
STEM CELL PRODUCT GRAM POSITIVE (Infections and infestations) | 1 (1) | 0 (0)
URINARY TRACT INFECTION (Infections and infestations) | 0 (0) | 1 (2)
VAGINAL INFECTION (Infections and infestations) | 0 (0) | 1 (1)
VIRIDANS STREPTOCOCCI BACTEREMIA (Infections and infestations) | 0 (0) | 1 (1)
BRUISING (Injury, poisoning and procedural complications) | 10 (12) | 8 (8)
FALL (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
LIP LESION (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
SKIN EXCORIATION (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
ACTIVATED PARTIAL THROMBOPLASTIN TIME PROLONGED (Investigations) | 1 (1) | 2 (2)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 8 (9) | 7 (7)
ALKALINE PHOSPHATASE INCREASED (Investigations) | 6 (6) | 4 (4)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 8 (8) | 5 (5)
BLOOD BILIRUBIN INCREASED (Investigations) | 8 (9) | 1 (1)
CARDIAC TROPONIN I INCREASED (Investigations) | 2 (2) | 0 (0)
CREATININE INCREASED (Investigations) | 3 (3) | 3 (4)
ELECTROCARDIOGRAM QT CORRECTED INTERVAL PROLONGED (Investigations) | 2 (2) | 0 (0)
LYMPHOCYTE COUNT DECREASED (Investigations) | 19 (34) | 19 (32)
NEUTROPHIL COUNT DECREASED (Investigations) | 19 (27) | 17 (27)
PLATELET COUNT DECREASED (Investigations) | 18 (29) | 19 (34)
WEIGHT GAIN (Investigations) | 12 (13) | 4 (6)
WEIGHT LOSS (Investigations) | 6 (7) | 11 (13)
WHITE BLOOD CELL DECREASED (Investigations) | 18 (33) | 18 (34)
ALKALOSIS (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
ANOREXIA (Metabolism and nutrition disorders) | 16 (21) | 16 (20)
DEHYDRATION (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
HYPERCALCEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
HYPERGLYCEMIA (Metabolism and nutrition disorders) | 4 (5) | 3 (5)
HYPERKALEMIA (Metabolism and nutrition disorders) | 2 (2) | 2 (2)
HYPERMAGNESEMIA (Metabolism and nutrition disorders) | 2 (3) | 1 (1)
HYPERNATREMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
HYPERTRIGLYCERIDEMIA (Metabolism and nutrition disorders) | 7 (7) | 13 (13)
HYPERURICEMIA (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
HYPOALBUMINEMIA (Metabolism and nutrition disorders) | 18 (23) | 17 (23)
HYPOCALCEMIA (Metabolism and nutrition disorders) | 14 (16) | 10 (11)
HYPOGLYCEMIA (Metabolism and nutrition disorders) | 2 (4) | 4 (4)
HYPOKALEMIA (Metabolism and nutrition disorders) | 19 (28) | 18 (26)
HYPOMAGNESEMIA (Metabolism and nutrition disorders) | 19 (22) | 17 (19)
HYPONATREMIA (Metabolism and nutrition disorders) | 19 (29) | 19 (29)
HYPOPHOSPHATEMIA (Metabolism and nutrition disorders) | 14 (19) | 12 (12)
OBESITY (Metabolism and nutrition disorders) | 2 (2) | 3 (5)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 6 (7) | 4 (5)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 13 (13) | 9 (12)
BONE PAIN (Musculoskeletal and connective tissue disorders) | 6 (7) | 8 (11)
CHEST WALL PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
DYSTONIA (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
FLANK PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
GENERALIZED MUSCLE WEAKNESS (Musculoskeletal and connective tissue disorders) | 13 (17) | 10 (13)
HIP PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
MYALGIA (Musculoskeletal and connective tissue disorders) | 4 (4) | 3 (3)
MYOCLONIC JERKS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
NECK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 4 (5)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 11 (14) | 5 (6)
FOCAL INTRAMUCOSAL ADENOCARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
AMNESIA (Nervous system disorders) | 1 (1) | 0 (0)
COGNITIVE DISTURBANCE (Nervous system disorders) | 1 (1) | 3 (3)
CONCENTRATION IMPAIRMENT (Nervous system disorders) | 1 (1) | 0 (0)
DEPRESSED LEVEL OF CONSCIOUSNESS (Nervous system disorders) | 1 (1) | 0 (0)
DIZZINESS (Nervous system disorders) | 5 (5) | 5 (5)
DYSGEUSIA (Nervous system disorders) | 8 (8) | 5 (6)
DYSPHASIA (Nervous system disorders) | 0 (0) | 1 (1)
HEADACHE (Nervous system disorders) | 13 (17) | 16 (23)
HYPERSOMNIA (Nervous system disorders) | 1 (1) | 0 (0)
LETHARGY (Nervous system disorders) | 3 (3) | 2 (2)
MEMORY IMPAIRMENT (Nervous system disorders) | 1 (1) | 2 (2)
PARESTHESIA (Nervous system disorders) | 4 (5) | 4 (5)
PERIPHERAL SENSORY NEUROPATHY (Nervous system disorders) | 8 (10) | 4 (4)
PRESYNCOPE (Nervous system disorders) | 1 (1) | 0 (0)
SOMNOLENCE (Nervous system disorders) | 4 (4) | 2 (2)
SYNCOPE (Nervous system disorders) | 1 (1) | 0 (0)
TREMOR (Nervous system disorders) | 5 (5) | 0 (0)
AGGRAVATION (Psychiatric disorders) | 0 (0) | 1 (1)
AGITATION (Psychiatric disorders) | 5 (5) | 2 (2)
ANXIETY (Psychiatric disorders) | 10 (14) | 8 (10)
CONFUSION (Psychiatric disorders) | 4 (4) | 2 (2)
DELIRIUM (Psychiatric disorders) | 1 (1) | 0 (0)
DEPRESSION (Psychiatric disorders) | 2 (3) | 2 (2)
HALLUCINATIONS (Psychiatric disorders) | 2 (2) | 0 (0)
INSOMNIA (Psychiatric disorders) | 8 (8) | 10 (10)
RESTLESSNESS (Psychiatric disorders) | 4 (4) | 1 (1)
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 3 (3) | 0 (0)
ACUTE RENAL INSUFFICIENCY (Renal and urinary disorders) | 0 (0) | 1 (1)
BLADDER SPASM (Renal and urinary disorders) | 4 (4) | 0 (0)
BPH (Renal and urinary disorders) | 1 (1) | 0 (0)
CYSTITIS NONINFECTIVE (Renal and urinary disorders) | 2 (2) | 0 (0)
DYSURIA (Renal and urinary disorders) | 1 (1) | 0 (0)
HEMATURIA (Renal and urinary disorders) | 11 (11) | 7 (7)
PROTEINURIA (Renal and urinary disorders) | 9 (9) | 2 (2)
URINARY FREQUENCY (Renal and urinary disorders) | 6 (6) | 2 (2)
URINARY INCONTINENCE (Renal and urinary disorders) | 3 (3) | 0 (0)
URINARY RETENTION (Renal and urinary disorders) | 0 (0) | 1 (1)
URINARY TRACT PAIN (Renal and urinary disorders) | 4 (5) | 1 (1)
URINARY URGENCY (Renal and urinary disorders) | 2 (2) | 1 (1)
GENITAL EDEMA (Reproductive system and breast disorders) | 1 (1) | 0 (0)
MENORRHAGIA (Reproductive system and breast disorders) | 0 (0) | 1 (1)
PELVIC PAIN (Reproductive system and breast disorders) | 1 (1) | 0 (0)
PENILE PAIN (Reproductive system and breast disorders) | 1 (1) | 0 (0)
SCROTAL EDEMA (Reproductive system and breast disorders) | 1 (1) | 0 (0)
SCROTAL PAIN (Reproductive system and breast disorders) | 3 (3) | 0 (0)
VAGINAL DISCHARGE (Reproductive system and breast disorders) | 0 (0) | 1 (1)
VAGINAL DRYNESS (Reproductive system and breast disorders) | 0 (0) | 1 (1)
VAGINAL HEMORRHAGE (Reproductive system and breast disorders) | 0 (0) | 1 (1)
VAGINAL ITCH (Reproductive system and breast disorders) | 0 (0) | 1 (1)
VAGINAL PAIN (Reproductive system and breast disorders) | 0 (0) | 1 (1)
VAGINAL SORES (Reproductive system and breast disorders) | 0 (0) | 1 (1)
ALLERGIC RHINITIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
ASPIRATION (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
COUGH (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 7 (8)
DYSPNEA (Respiratory, thoracic and mediastinal disorders) | 7 (9) | 1 (1)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 5 (5)
HICCUPS (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3)
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 6 (8) | 3 (3)
LUNG CRACKLES (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 5 (5)
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 5 (6) | 0 (0)
POSTNASAL DRIP (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
PRODUCTIVE COUGH (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
PULMONARY EDEMA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
PULOMONARY NODULES (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
SENSITIVITY TO SMELL (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
SLEEP APNEA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
SNEEZING (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
SORE THROAT (Respiratory, thoracic and mediastinal disorders) | 6 (7) | 9 (10)
VOICE ALTERATION (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
WHEEZING (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
ALLERGIC DERMITIS (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
BULLOUS DERMATITIS (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
DRY SKIN (Skin and subcutaneous tissue disorders) | 5 (5) | 10 (12)
ECZEMA (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
ERYTHEMA TOE (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
FOLLICULAR SKIN LESIONS (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
HICKMAN CATHETER EXIT SITE REDNESS (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
HICKMAN SITE INFLAMMATION (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
L ANKLE LACERATION (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
L THIGH TUMOR (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
LEFT TOE INFLAMMATION (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
PALLOR (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
PALMARPLANTAR ERYTHRODYSESTHESIA SYNDROME (Skin and subcutaneous tissue disorders) | 2 (2) | 4 (4)
PERIORBITAL EDEMA (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
PRURITUS (Skin and subcutaneous tissue disorders) | 7 (8) | 10 (11)
RASH ACNEIFORM (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3)
RASH MACULOPAPULAR (Skin and subcutaneous tissue disorders) | 10 (10) | 11 (12)
RED SPOTS ON CALVES (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
SCALP PAIN (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
SKIN ABRASION (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
SKIN HYPERPIGMENTATION (Skin and subcutaneous tissue disorders) | 4 (4) | 6 (6)
SKIN ULCERATION (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
URTICARIA (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
FLUSHING (Vascular disorders) | 7 (7) | 5 (5)
HEMATOMA (Vascular disorders) | 1 (1) | 0 (0)
HYPERTENSION (Vascular disorders) | 17 (32) | 17 (23)
HYPOTENSION (Vascular disorders) | 11 (13) | 9 (13)
SUPERFICIAL THROMBOPHLEBITIS (Vascular disorders) | 1 (1) | 0 (0)
VASCULAR CONGESTION (Vascular disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-07-03): https://cdn.clinicaltrials.gov/large-docs/59/NCT03128359/Prot_SAP_000.pdf